CLINICAL TRIAL: NCT02720796
Title: A Prospective Correlative Trial of Personalized Patient-Derived Xenograft (PDX or TumorGraft) Modeling in Adult Patients With Metastatic or Recurrent Sarcoma
Brief Title: Patient-Derived Xenograft (PDX) Modeling in Adult Patients With Metastatic or Recurrent Sarcoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment barriers
Sponsor: Champions Oncology (Industry)
Collaborators: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CO-001
Record Dates: First submitted 2015-11-05; First posted 2016-03-28 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Sarcoma
Keywords: PDX; TumorGraft; Patient derived xenograft; sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PDX drug sensitivity testing (Other): Patient derived xenograft (PDX) models will be developed for each patient and drug activity assessed in their personalized PDX model. PDX drug sensitivity information will be provided to the treating physician.
  Interventions: Other: PDX drug sensitivity testing

INTERVENTIONS:
Other: PDX drug sensitivity testing — Patient derived xenograft (PDX) models will be developed for each patient and drug activity assessed in their personalized PDX model. PDX drug sensitivity information will be provided to the treating physician.

SUMMARY:
Patients with recurrent or metastatic sarcoma will be consented to develop a patient derived xenograft (PDX or TumorGraft) model of their tumor to perform drug sensitivity testing. The purpose of the study is to evaluate the accuracy of the patient derived xenograft (PDX) model in predicting patient clinical response to the same drug treatment.

ELIGIBILITY:
* 15 years of age or older
* Patients with metastatic sarcoma who have had no more than one prior systemic treatment for metastatic disease
* Patients with recurrent sarcoma at relapse
* Patients with confirmed histological diagnosis of sarcoma or suspected diagnosis of sarcoma. Some specific subtypes of sarcoma are NOT eligible (Gastrointestinal Stromal Tumor (GIST), carcinosarcoma, sarcomatoid mesothelioma, and metastatic phyllodes tumor)
* If initial suspected diagnosis of sarcoma, must have sarcoma diagnosis confirmed prior to proceeding with PDX drug sensitivity testing
* Must have measureable disease for computed tomography (CT) scan or magnetic resonance imaging (MRI) evaluation following biopsy or surgery to obtain tissue for PDX development.
* No plan for concurrent chemoradiation, for target lesions that will be used for drug treatment correlation with PDX
* Fresh tumor tissue available for PDX development
* Eastern Cooperative Oncology Group performance status of 0-1
* Life expectancy exceeds 6 months
* Plan to receive systemic therapy
* Informed consent

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-11; Primary Completion 2017-11-30 (Estimated); Study Completion 2017-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients' whose personalized PDX model accurately predicts clinical response to therapy with same drug treatment. | 3 years
  Overall accuracy as assessed by evaluating Response Evaluation Criteria In Solid Tumors (RECIST) criteria in patient tumor and correlating to tumor regression in PDX model for same drug treatment.

SECONDARY OUTCOMES:
Number of patients' whose personalized PDX model accurately predicts clinical response to therapy over subsequent lines of therapy. | 3 years
  Overall accuracy as assessed by evaluating RECIST criteria in patient and correlating to tumor regression in PDX model for same drug treatment, over subsequent lines of therapy.
Factors that impact on engraftment success. | 2 years
  % engraftment of tumor as a function of patient and tumor characteristics.
Factors that impact time to drug sensitivity testing. | 2 years
  Time to PDX drug sensitivity testing as a function of patient and tumor characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Albiruni Razak, MD, Principal Investigator — Mount Sinai Hospital, Toronto, Ontario, Canada
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada